CLINICAL TRIAL: NCT04252300
Title: Open Label, Fixed Sequences, One-way Cross-over Study to Determine the Effects of Multiple Doses BAY1817080 (150 mg) on the Pharmacokinetics of a 5 mg Dose Rosuvastatin in Healthy Participants
Brief Title: Study to Learn the Effect of Drug BAY1817080 on the Way the Body Absorbs, Distributes and Excretes Another Drug Rosuvastatin in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20246
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Drug Interactions
Keywords: P2X3 receptor antagonist; Rosuvastatin; Organic Anion Transporting Polypeptide 1B1 (OATP1B1); Organic Anion Transporting Polypeptide 1B3 (OATP1B3); Breast Cancer Resistance Protein (BCRP); Pain; Chronic cough; Cholesterol
MeSH Terms: conditions — Pain; Chronic Cough | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Healthy subjects_Period 1 (Experimental): Healthy adults from USA receive a single dose of rosuvastatin (interaction drug) in Period 1.
  Interventions: Drug: Rosuvastatin
- Healthy subjects_Period 2 (Experimental): The healthy adults from Period 1 receive both rosuvastatin + BAY1817080 in Period 2.
  Interventions: Drug: Rosuvastatin + BAY1817080

INTERVENTIONS:
Drug: Rosuvastatin — Single dose of 5 mg rosuvastatin is administered as tablet orally on Day 1 of Period 1 (total length = 5 days).
  Other Names: Crestor®
  Arms: Healthy subjects_Period 1
Drug: Rosuvastatin + BAY1817080 — A single dose of 5 mg rosuvastatin tablets is administered on Day 8 of Period 2 (total length = 15 days). BAY1817080 is administered as tablets twice daily on Days 1 to 14 of Period 2.
  Other Names: P2X3 receptor antagonist;; Crestor®
  Arms: Healthy subjects_Period 2

SUMMARY:
Researchers in this study want to learn how the study drug BAY1817080 interacts with another drug called rosuvastatin (brand name: Crestor) and affects the way the body absorbs, distributes and excretes rosuvastatin in healthy adult male and female participants (drug-drug interaction study). The study drug BAY1817080 is a new drug under development with a goal to suppress pain and chronic cough. It works by binding to and blocking proteins related to pain in the body. Rosuvastatin is an approved and marketed drug to lower high levels of "bad" cholesterol (a waxy, fat-like substance found in blood). Both drugs interact with the same proteins (molecules) in the human body, and as a result, the study drug may affect the way rosuvastatin is taken up and used by the body when applied together.

Participants in this study will be asked to visit the clinic 3 times over a period of 3 to 4 weeks. Each participant will receive rosuvastatin tablets twice with at least 11 days in between and the study drug tablets twice daily for 14 days. Blood samples will be taken from the participants to measure the blood levels of rosuvastatin.

DETAILED DESCRIPTION:
The primary objective of the study is to investigate the influence of multiple doses of BAY1817080 on the pharmacokinetics of rosuvastatin given concomitantly. Secondary objective is to investigate the safety of BAY1817080.

ELIGIBILITY:
Inclusion Criteria:

* Participant is healthy as determined by the investigator
* White or Black race
* Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m² at screening
* Body weight of at least 50 kg at screening

Exclusion Criteria:

* Known or suspected allergy or hypersensitivity to BAY1817080, rosuvastatin or any of their excipients
* Asian race
* Contraindications to rosuvastatin
* Any use of systemic or topically active medication or herbal remedies, prescription or non-prescription, within 1 week prior to the first study intervention administration or during the study until follow-up (occasional use of ibuprofen is permissible)
* History of or positive COVID-19 test or contact with COVID-19 positive subject in past 4 weeks

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-08-29 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration of rosuvastatin without concomitant administration of BAY1817080 (Cmax) | Predose and up to 15 hours after drug on Day 1, 0 and 12 hours on Day 2, 0 hours on Day 3, 4 and 5 of Period 1
Maximum plasma concentration of rosuvastatin after concomitant administration of BAY1817080 (Cmax1) | Predose and up to 15 hours after rosuvastatin on Day 8, 0 and 12 hours on Day 9, 0 hour on Days 10, 11, 12, 13, 14 and 15 of Period 2
Area under the concentration-time curve of rosuvastatin without concomitant administration of BAY1817080 (AUC) | Predose and up to 15 hours after drug on Day 1, 0 and 12 hours on Day 2, 0 hours on Day 3, 4 and 5 of Period 1
Area under the concentration-time curve of rosuvastatin after concomitant administration of BAY1817080 (AUC1) | Predose and up to 15 hours after rosuvastatin on Day 8, 0 and 12 hours on Day 9, 0 hour on Days 10, 11, 12, 13, 14 and 15 of Period 2

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Up to 10 weeks
Severity of treatment-emergent adverse events | Up to 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit, Inc., Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.